CLINICAL TRIAL: NCT00459758
Title: Pilot Study Using Electrical Stimulation on Hypertension
Brief Title: Effect of Electrical Stimulation at Acupoints on Blood Pressure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD0922060043
Record Dates: First submitted 2007-04-10; First posted 2007-04-12 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2007-07

CONDITIONS: Hypertension
Keywords: hypertension; Hans; Electrical stimulation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Hans unit

SUMMARY:
To determine if electrical stimulation on acupoints has any effect on hypertensive subjects.

DETAILED DESCRIPTION:
All subjects will be assigned into control and experimental groups by a random table. The first 40 numbers in the first row will be used for the study. Subjects assigned with an odd number will be divided into the control group.

ROLE OF SUBJECTS Subjects in the experimental will receive Hans treatment for hypertension. No invasive procedures will be used for subjects in either the control and experimental groups.

This randomized controlled study will recruit hypertensive subjects into control and experimental groups using a random table. Only the subjects in the experimental group use Hans stimulation as a treatment for high blood pressure. The treatment regiment is discussed in the Treatment section in detail. The subjects in the control group will not

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild hypertension (160-140/100-90 mmHg), male and female subjects with any racial background will be invited to participate in the study.
* All adult age groups are included in the study.
* Subjects must sign an informed consent form.

Exclusion Criteria:

* Diagnosis of severe hypertension (200-161/120-101 mmHg), limited physical activity, heart failure, kidney diseases and mental diseases are excluded in the study. A questionnaire will be used in the initial patient screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-01; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Blood pressure measurements.

CONTACTS AND LOCATIONS:
Overall Officials: John Zhang, MD, PhD, Principal Investigator — Logan University
Locations (1):
- Logan University, Chesterfield, Missouri, United States